CLINICAL TRIAL: NCT05507580
Title: A Phase 3b/4 Randomized, Blinded, Treat-to-Target and Dose-Flexibility Study of Upadacitinib in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Assess Treat-to-Target and Dosing Flexibility of Oral Upadacitinib Tablets in Adult Participants With Moderate to Severe Atopic Dermatitis
Acronym: Flex-Up
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-000; 2022-000434-42 (EudraCT Number)
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis (AD); Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- UPA 15 mg Double-Blind Treatment Period (Experimental): Participants received 15 mg upadacitinib orally once daily (QD) for 12 weeks during the Double-Blind Treatment Period.
  Interventions: Drug: Upadacitinib
- UPA 30 mg Double-Blind Treatment Period (Experimental): Participants received 30 mg upadacitinib orally once daily (QD) for 12 weeks during the Double-Blind Treatment Period.
  Interventions: Drug: Upadacitinib
- UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (Experimental): At Week 12 in the Double-Blind Treatment Period, participants receiving 15 mg upadacitinib orally once daily (QD) achieving a ≥ 90% reduction in the Eczema Area and Severity Index (EASI) (≥ EASI 90) were allocated to receive 15 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
  Interventions: Drug: Upadacitinib
- UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (Experimental): At Week 12 in the Double-Blind Treatment Period, participants receiving 15 mg upadacitinib orally once daily (QD) achieving a < 90% reduction in the Eczema Area and Severity Index (EASI) (< EASI 90) were allocated to receive 30 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
  Interventions: Drug: Upadacitinib
- UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (Experimental): At Week 12 in the Double-Blind Treatment Period, participants receiving 30 mg upadacitinib orally once daily (QD) achieving a ≥ 90% reduction in the Eczema Area and Severity Index (EASI) (≥ EASI 90) were allocated to receive 15 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
  Interventions: Drug: Upadacitinib
- UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (Experimental): At Week 12 in the Double-Blind Treatment Period, participants receiving 30 mg upadacitinib orally once daily (QD) achieving a < 90% reduction in the Eczema Area and Severity Index (EASI) (< EASI 90) were allocated to receive 30 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral tablet
  Other Names: RINVOQ; ABT-494

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Therapies spread over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study evaluates the dosing flexibility of upadacitinib in adult participants with moderate to severe AD. Adverse events and change in the disease activity will be assessed.

Upadacitinib is an approved drug for the treatment of moderate to severe/active immune-mediated inflammatory diseases such as rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, ulcerative colitis (UC), Crohn's Disease (CD), and AD. The study is comprised of a 35-day Screening Period, a 12-week double-blind period and a 12-week single-blind period. During the double-blind period, participants are placed in 1 of 2 groups, called treatment arms and will be randomized in a 1:1 ratio to receive upadacitinib. At 12 weeks during the single blind period, participants will be blinded to the upadacitinib dose based on their EASI response and reassigned to in 1 of 4 arms. After the last study visit, there is a 30-day follow-up visit. Approximately 454 adult participants ages 18 to 64 with moderate to severe AD who are candidates for systemic therapy will be enrolled at up to 160 sites worldwide.

The study is comprised of a 12-week double-blind period, followed by a 12-week single-blind period. Participants will receive upadacitinib oral tablets once daily for up to 24 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atopic dermatitis (AD) with onset of symptoms at least 3 years prior to Baseline and participant meets Hanifin and Rajka criteria.
* Eczema Area and Severity Index (EASI) score >= 16, vIGA-AD score >= 3 and >= 10% Body Surface Area (BSA) of AD involvement at the Baseline Visit.
* Baseline weekly average of daily Worst Pruritus NRS >= 4.
* Candidate for systemic treatment defined as prior use of systemic treatment for AD, OR previous inadequate response to TCS, TCI or PDE-4 inhibitors, OR for whom topical treatments are otherwise medically inadvisable.

Exclusion Criteria:

* Participants with current or past history of infection including:

  * Two or more episodes of herpes zoster, or one or more episodes of disseminated herpes zoster;
  * One or more episodes of disseminated herpes simplex (including eczema herpeticum);
  * Human immunodeficiency virus (HIV) infection defined as confirmed positive anti-HIV antibody (HIV Ab) test;
  * Active tuberculosis (TB) or meet TB exclusionary parameters (protocol specified requirements for TB testing);
  * Japan only: Positive result of beta-D-glucan (screening for Pneumocystis jirovecii infection) or two consecutive indeterminate results of beta-D-glucan during the Screening Period;
  * Active infection(s) requiring treatment with intravenous anti-infectives within 30 days, or oral/intramuscular anti-infectives within 14 days prior to the Baseline Visit;
  * Chronic recurring infection and/or active viral infection that, based on the investigator's clinical assessment, makes the participant an unsuitable candidate for the study;
  * COVID-19 infection: In participants who tested positive for COVID, at least 5 days must have passed since a COVID-19 positive test result for study entry of asymptomatic participants. Participants with mild/moderate COVID-19 infection can be enrolled if fever is resolved without use of antipyretics for 24 hours and other symptoms improved, or if 5 days have passed since the COVID-19 positive test result (whichever comes last). Participants may be rescreened if judged to be in good general health, as determined by the investigator based upon the medical history and physical examination.
* Evidence of Hepatitis B virus (HBV) or Hepatitis C virus (HCV).
* Any of the following medical diseases or disorders:

  * Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting, and aorto-coronary bypass surgery;
  * History of an organ transplant which requires continued immunosuppression;
  * History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class;
  * History of gastrointestinal perforation (other than due to appendicitis or mechanical injury), diverticulitis, or significantly increased risk for gastrointestinal perforation per investigator judgment;
  * Conditions that could interfere with drug absorption including but not limited to short bowel syndrome or gastric bypass surgery; participants with a history of gastric banding/segmentation are not excluded;
  * History of malignancy except for successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 461 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (106):
- Australia (5):
  - Momentum Clinical Research /ID# 254028, Darlinghurst, New South Wales
  - Premier Specialist /ID# 246150, Kogarah, New South Wales
  - Veracity Clinical Research /ID# 246154, Woolloongabba, Queensland
  - North Eastern Health Specialists /ID# 246153, Campbelltown, South Australia
  - Skin Health Institute Inc /ID# 246146, Carlton, Victoria
- Belgium (5):
  - Cliniques Universitaires UCL Saint-Luc /ID# 245842, Woluwe-Saint-Lambert, Brussels Capital
  - Grand Hôpital De Charleroi - Notre Dame /ID# 245837, Charleroi, Hainaut
  - AZ Sint-Lucas /ID# 253708, Ghent, Oost-Vlaanderen
  - Dermatologie Maldegem /ID# 245840, Maldegem, Oost-Vlaanderen
  - CHU de Liege /ID# 245839, Liège
- Bulgaria (6):
  - UMHAT Alexandrovska EAD /ID# 246594, Sofiya, Sofia
  - Medical center Cordis /ID# 253310, Pleven
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 246395, Sofia
  - Ambulatory for Specialized Medical Care for skin and venereal diseases /ID# 247027, Sofia
  - Medical Center Euroderma /ID# 246736, Sofia
  - Medical center EuroHealth /ID# 246305, Sofia
- Canada (8):
  - Dermatology Research Institute - Blackfoot Trail /ID# 246703, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 246705, Calgary, Alberta
  - Rejuvenation Dermatology - Edmonton Downtown /ID# 256790, Edmonton, Alberta
  - Alberta DermaSurgery Centre /ID# 247286, Edmonton, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 246700, Surrey, British Columbia
  - Lynde Institute for Dermatology /ID# 246699, Markham, Ontario
  - SKiN Centre for Dermatology /ID# 246702, Peterborough, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 246698, Waterloo, Ontario
- China (5):
  - Beijing Friendship Hospital /ID# 247719, Beijing, Beijing Municipality
  - Peking University Third Hospital /ID# 247842, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University /ID# 247951, Guangzhou, Guangdong
  - The First Hospital of China Medical University /ID# 247686, Shenyang, Liaoning
  - Huashan Hospital, Fudan University /ID# 247680, Shanghai, Shanghai Municipality
- Germany (12):
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 245629, Blankenfelde-Mahlow, Brandenburg
  - Klinikum Darmstadt /ID# 247028, Darmstadt, Hesse
  - Universitaetsklinikum Frankfurt /ID# 245627, Frankfurt am Main, Hesse
  - Fachklinik Bad Bentheim /ID# 245634, Bad Bentheim, Lower Saxony
  - Studienzentrum an der Hase GbR Dr. Weyergraf/Dr. Frick/Thomas Heiber /ID# 245636, Bramsche, Lower Saxony
  - Universitaetsklinikum Muenster /ID# 245623, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus Dresden /ID# 248413, Dresden, Saxony
  - Elbe Klinikum Buxtehude /ID# 245626, Buxtehude
  - Derma Study Center Friedrichshafen GmbH /ID# 245640, Friedrichshafen
  - Universitaetsklinikum Halle (Saale) /ID# 245637, Halle
  - Dermatologikum Hamburg /ID# 245635, Hamburg
  - Dermatologie Quist-BAG Dres. med. Quist PartG /ID# 245628, Mainz
- Hungary (4):
  - Gyongyosi Bugat Pal Korhaz /ID# 246422, Gyöngyös, Heves County
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 246428, Kaposvár, Somogy County
  - Clinexpert Kft /ID# 246427, Budapest
  - DERMA-B Egeszsegugyi es Szolgaltato - Debrecen - Gyepusor Utca /ID# 246426, Debrecen
- Italy (6):
  - IRCCS Istituto Clinico Humanitas /ID# 246630, Rozzano, Lombardy
  - Duplicate_Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 254355, Ancona
  - Duplicate_ASST Spedali civili di Brescia /ID# 246631, Brescia
  - Universita degli Studi Gabriele dAnnunzio /ID# 246629, Chieti
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 246634, Milan
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 246632, Perugia
- Japan (6):
  - Miyata Dermatology Clinic /ID# 255491, Matsudo-Shi, Chiba
  - Fukuoka University Hospital /ID# 255182, Fukuoka, Fukuoka
  - Takagi Dermatological Clinic /ID# 255181, Obihiro-shi, Hokkaido
  - Nomura Dermatology Clinic /ID# 255534, Yokohama, Kanagawa
  - Tohoku University Hospital /ID# 255183, Sendai, Miyagi
  - Maruyama Dermatology Clinic /ID# 255441, Koto-ku, Tokyo
- Netherlands (2):
  - Amphia Ziekenhuis /ID# 246397, Breda, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 245673, Amsterdam, North Holland
- New Zealand (3):
  - Greenlane Clinical Centre /ID# 246556, Epsom, Auckland
  - Clinical Trials New Zealand /ID# 246557, Hamilton, Waikato Region
  - Aotearoa Clinical Trials /ID# 246559, Auckland
- Poland (13):
  - Duplicate_Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej Alergologia Plus /ID# 253508, Poznan, Greater Poland Voivodeship
  - Specjalistyczna Przychodnia Lekarska Alergo-Med sp. z o.o. /ID# 253846, Poznan, Greater Poland Voivodeship
  - Oftalmika sp. z o.o. /ID# 253429, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun /ID# 245749, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o. /ID# 245836, Krakow, Lesser Poland Voivodeship
  - CenterMed Krakow Sp. z o.o. /ID# 253940, Krakow, Lesser Poland Voivodeship
  - Klinika Ambroziak Sp. z o.o. /ID# 245748, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka /ID# 245746, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o. /ID# 245741, Gdansk, Pomeranian Voivodeship
  - Centrum Medyczne Pratia Gdynia /ID# 245835, Gdynia, Pomeranian Voivodeship
  - Silmedic Sp. z o.o. /ID# 253863, Katowice, Silesian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 246329, Lodz, Łódź Voivodeship
  - Santa Sp. z o.o. Santa Familia Centrum Badan, Profilaktyki i Leczenia /ID# 253872, Lodz, Łódź Voivodeship
- Portugal (4):
  - Centro Hospitalar de Lisboa Central /ID# 246247, Lisbon
  - Hospital CUF Descobertas /ID# 245702, Lisbon
  - Centro Hospitalar Universitario do Porto, EPE - Hospital Santo Antonio /ID# 245701, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 245704, Porto
- Slovakia (3):
  - Poliklinika Bezrucova (Cliniq s.r.o.) /ID# 247515, Bratislava
  - BeneDerma s.r.o. /ID# 247513, Bratislava
  - Univerzitna nemocnica Martin /ID# 246948, Martin, Žilina Region
- South Korea (6):
  - Korea University Ansan Hospital /ID# 245653, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 245654, Bucheon-si, Gyeonggido
  - Ajou University Hospital /ID# 245652, Suwon, Gyeonggido
  - Chungang University Hospital /ID# 245655, Dongjak-gu, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 245651, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 245657, Seoul, Seoul Teugbyeolsi
- Spain (8):
  - Hospital Universitario Germans Trias i Pujol /ID# 246320, Badalona, Barcelona
  - Hospital Universitari de Bellvitge /ID# 246326, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 253820, Majadahonda, Madrid
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 246270, Alicante
  - Hospital Universitario Infanta Leonor /ID# 246272, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 246273, Madrid
  - Complejo Hospitalario Universitario de Pontevedra /ID# 246323, Pontevedra
  - Hospital Universitario Virgen del Rocio /ID# 253822, Seville
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 245710, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 245711, Taipei City, Taipei
  - Chung Shan Medical University Hospital /ID# 245707, Taichung
  - Mackay Memorial Hospital /ID# 245713, Taipei
  - Taipei Municipal Wan Fang Hospital /ID# 245712, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 245709, Taoyuan
- United Kingdom (4):
  - University Hospital Southampton NHS Foundation Trust /ID# 246393, Southampton, Hampshire
  - NHS Greater Glasgow and Clyde /ID# 246253, Glasgow, Scotland
  - Leeds Teaching Hospitals NHS Trust /ID# 246241, Leeds, West Yorkshire
  - NHS Lothian /ID# 246245, Edinburgh

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised of a 35-day Screening Period, a 12-week Double-Blind Treatment Period and a 12-week Single-Blind Treatment Period. During the Single-Blind Period, participants were blinded to the upadacitinib dose and Eczema Area and Severity Index (EASI) score evaluations.
Period: Double-Blind Treatment Period
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Started | 229 | 232 | 0 | 0 | 0 | 0
Completed | 217 | 226 | 0 | 0 | 0 | 0
Not Completed | 12 | 6 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 1 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 5 | 4 | 0 | 0 | 0 | 0
Period: Single-Blind Treatment Period
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Started | 0 | 0 | 72 | 144 | 133 | 91
Completed | 0 | 0 | 70 | 132 | 126 | 79
Not Completed | 0 | 0 | 2 | 12 | 7 | 12
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 5 | 2 | 6
Not completed — Other, not specified | 0 | 0 | 2 | 7 | 3 | 5

BASELINE CHARACTERISTICS:
Population: ITT_1 Population: all participants who were randomized in the Double-Blind Treatment Period
Groups:
- Total: Total of all reporting groups
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period | Total
Number analyzed (Participants) | 229 | 232 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.4 (12.06) | 32.7 (10.83) | 33.5 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 110 | 205
  Male | 134 | 122 | 256
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 219 | 223 | 442
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 67 | 66 | 133
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 2 | 3 | 5
  White | 155 | 158 | 313
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) at Week 24
Description: The EASI is a composite index with scores ranging from 0 to 72. Four atopic dermatitis (AD) disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are assessed for severity on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%).
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT_2) Population: all participants who were allocated to an assigned dose at Week 12 for the Single-Blind Treatment Period; participants with available data, as observed analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 71 | 133 | 130 | 82
percentage of participants | 74.6 [64.5 to 84.8] | 48.1 [39.6 to 56.6] | 68.5 [60.5 to 76.4] | 29.3 [19.4 to 39.1]

2. Secondary Outcome: Percentage of Participants Achieving ≥ 75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 75) at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 71 | 133 | 130 | 82
percentage of participants | 97.2 [93.3 to 100.0] | 69.2 [61.3 to 77.0] | 88.5 [83.0 to 94.0] | 52.4 [41.6 to 63.2]

3. Secondary Outcome: Percentage of Participants Achieving a 100% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 100) at Week 24
Description: as for outcome 1
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 71 | 133 | 130 | 82
percentage of participants | 33.8 [22.8 to 44.8] | 7.5 [3.0 to 12.0] | 21.5 [14.5 to 28.6] | 3.7 [0.0 to 7.7]

4. Secondary Outcome: Percentage of Participants Achieving ≥ 75% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 75) at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT_1) Population: all participants who were randomized in the Double-Blind Treatment Period; participants with available data, as observed analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 222 | 227
percentage of participants | 64.4 [58.1 to 70.7] | 79.3 [74.0 to 84.6]

5. Secondary Outcome: Percentage of Participants Achieving ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 222 | 227
percentage of participants | 33.8 [27.6 to 40.0] | 59.9 [53.5 to 66.3]

6. Secondary Outcome: Percentage of Participants Achieving a 100% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 100) at Week 12
Description: as for outcome 1
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 222 | 227
percentage of participants | 7.7 [4.2 to 11.2] | 15.9 [11.1 to 20.6]

7. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) and Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 12 Among Those With WP-NRS > 1 at Baseline
Description: The EASI is a composite index with scores ranging from 0 to 72. Four atopic dermatitis (AD) disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) assessed for severity on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%).
  The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants rated itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 183 | 194
percentage of participants | 18.0 [12.5 to 23.6] | 32.5 [25.9 to 39.1]

8. Secondary Outcome: Percentage of Participants Achieving a ≥ 90% Reduction From Baseline in Eczema Area and Severity Index Score (EASI 90) and Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) at Week 24 Among Those With WP-NRS > 1 at Baseline
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 52 | 82 | 100 | 59
percentage of participants | 38.5 [25.2 to 51.7] | 20.7 [12.0 to 29.5] | 35.0 [25.7 to 44.3] | 20.3 [10.1 to 30.6]

9. Secondary Outcome: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vlGA-AD) of 0 or 1 at Week 12
Description: vIGA-AD is a validated assessment instrument used in clinical studies to rate the severity of AD globally. A 5-point scale is used to measure the severity of disease at the time of the investigator's evaluation of the participant ranging from 0 - Clear (no inflammatory signs of atopic dermatitis [no erythema, no induration/papulation, no lichenification, no oozing/crusting] Post-inflammatory hyperpigmentation and/or hypopigmentation may be present) to 4 - Severe (marked erythema [deep or bright red], marked induration/papulation, and/or marked lichenification).
Time Frame: At Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 222 | 227
percentage of participants | 29.7 [23.7 to 35.7] | 51.5 [45.0 to 58.0]

10. Secondary Outcome: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vlGA-AD) of 0 or 1 at Week 24
Description: as for outcome 9
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period: At Week 12 in the Double-Blind Treatment Period, participants receiving 15 mg upadacitinib orally once daily (QD) achieving a ≥90% reduction in the Eczema Area and Severity Index (EASI) (≥EASI 90) were allocated to receive 15 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
- UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period: At Week 12 in the Double-Blind Treatment Period, participants receiving 30 mg upadacitinib orally once daily (QD) achieving a ≥90% reduction in the Eczema Area and Severity Index (EASI) (≥EASI 90) were allocated to receive 15 mg upadacitinib orally once daily (QD) for 12 weeks during the Single-Blind Treatment Period.
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 71 | 133 | 130 | 82
percentage of participants | 63.4 [52.2 to 74.6] | 40.6 [32.3 to 48.9] | 52.3 [43.7 to 60.9] | 29.3 [19.4 to 39.1]

11. Secondary Outcome: Percentage of Participants Achieving an Improvement (Reduction) in Worst Pruritus Numerical Rating Scale (WP-NRS) ≥4 at Week 12 Among Those With Baseline WP-NRS ≥4
Description: The Worst Pruritus NRS is an assessment tool that participants used to report the intensity of their pruritus during a 24-hour recall period using an electronic hand-held device. Participants rated itch (pruritus) intensity at its worst during the past 24 hours on an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 182 | 195
percentage of participants | 53.3 [46.0 to 60.5] | 67.7 [61.1 to 74.3]

12. Secondary Outcome: Percentage of Participants Achieving an Improvement (Reduction) in Worst Pruritus Numerical Rating Scale (WP-NRS) ≥4 at Week 24 Among Those With Baseline WP-NRS ≥4
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 52 | 82 | 100 | 60
percentage of participants | 73.1 [61.0 to 85.1] | 57.3 [46.6 to 68.0] | 67.0 [57.8 to 76.2] | 60.0 [47.6 to 72.4]

13. Secondary Outcome: Percentage of Participants Achieving Worst Pruritus Numerical Rating Scale (WP-NRS) of 0 or 1 at Week 12 Among Those With Baseline WP-NRS >1
Description: as for outcome 11
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 183 | 195
percentage of participants | 27.3 [20.9 to 33.8] | 40.0 [33.1 to 46.9]

14. Secondary Outcome: Percentage of Participants Achieving Worst Pruritus Numerical Rating Scale (WP-NRS) of 0 or 1 at Week 24 Among Those With Baseline WP-NRS >1
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 52 | 83 | 100 | 60
percentage of participants | 46.2 [32.6 to 59.7] | 32.5 [22.5 to 42.6] | 38.0 [28.5 to 47.5] | 28.3 [16.9 to 39.7]

15. Secondary Outcome: Percentage of Participants Achieving Improvement (Reduction) in Dermatology Life Quality Index (DLQI) ≥4 at Week 12 Among Those With Baseline DLQI ≥4
Description: DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of atopic dermatitis (AD) disease symptoms and treatment on health-related quality of life (HRQoL). It consists of 10 questions assessing impact of skin diseases on different aspects of participant's QoL over the prior week. Each item is scored on a 4-point scale: 0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much. Item scores (0 to 3) are added to provide a total score range of 0 to 30. Higher scores indicate greater impairment of HRQoL.
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 213 | 216
percentage of participants | 77.5 [71.9 to 83.1] | 88.9 [84.7 to 93.1]

16. Secondary Outcome: Percentage of Participants Achieving Improvement (Reduction) in Dermatology Life Quality Index (DLQI) ≥4 at Week 24 Among Those With Baseline DLQI ≥4
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 67 | 129 | 124 | 77
percentage of participants | 88.1 [80.3 to 95.8] | 82.2 [75.6 to 88.8] | 84.7 [78.3 to 91.0] | 74.0 [64.2 to 83.8]

17. Secondary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) of 0 or 1 At Week 12 Among Those With Baseline DLQI >1
Description: as for outcome 15
Time Frame: Baseline and Week 12
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period
Number analyzed (Participants) | 216 | 222
percentage of participants | 22.2 [16.7 to 27.8] | 36.5 [30.2 to 42.8]

18. Secondary Outcome: Percentage of Participants Achieving Dermatology Life Quality Index (DLQI) of 0 or 1 At Week 24 Among Those With Baseline DLQI >1
Description: as for outcome 15
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
Number analyzed (Participants) | 69 | 129 | 127 | 79
percentage of participants | 42.0 [30.4 to 53.7] | 24.0 [16.7 to 31.4] | 35.4 [27.1 to 43.8] | 15.2 [7.3 to 23.1]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time informed consent was signed to the end of the study. The median time on follow-up was 168 days for the Double-Blind Treatment Period groups and ranged from 168 to 169 days for the Single-Blind Treatment Period groups.
Arm/Group | UPA 15 mg Double-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period
All-Cause Mortality (participants affected / at risk) | 0/229 | 0/232 | 0/72 | 0/144 | 0/133 | 0/91
Serious Adverse Events (participants affected / at risk) | 8/229 | 0/232 | 1/72 | 1/144 | 1/133 | 0/91
Other Adverse Events (participants affected / at risk) | 41/229 | 67/232 | 17/72 | 38/144 | 39/133 | 33/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UPA 15 mg Double-Blind Treatment Period (N=229) | UPA 30 mg Double-Blind Treatment Period (N=232) | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (N=72) | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (N=144) | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (N=133) | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (N=91)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXIC NODULAR GOITRE (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPIDIDYMITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UPA 15 mg Double-Blind Treatment Period (N=229) | UPA 30 mg Double-Blind Treatment Period (N=232) | UPA 15 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (N=72) | UPA 15 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (N=144) | UPA 30 mg Double-Blind Treatment Period --> UPA 15 mg Single-Blind Treatment Period (N=133) | UPA 30 mg Double-Blind Treatment Period --> UPA 30 mg Single-Blind Treatment Period (N=91)
NASOPHARYNGITIS (Infections and infestations) | 13 (17) | 21 (24) | 8 (9) | 6 (7) | 10 (11) | 2 (2)
ORAL HERPES (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 9 (11) | 5 (5) | 3 (3) | 4 (5) | 4 (4)
ACNE (Skin and subcutaneous tissue disorders) | 16 (16) | 32 (32) | 1 (1) | 4 (4) | 8 (8) | 6 (6)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 7 (7) | 9 (10) | 6 (6) | 23 (24) | 16 (17) | 15 (15)
ECZEMA (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT05507580/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT05507580/SAP_001.pdf